CLINICAL TRIAL: NCT01694992
Title: Randomized Clinical Trial of Very Early Rehabilitation Compared With Conventional Rehabilitation in Acute Ischemic Stroke in the Vascular Unit of the Hospital de Clínicas de Porto Alegre - HCPA
Brief Title: Very Early Rehabilitation in Acute Ischemic Stroke
Acronym: VERIS-Brazil
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11.0121
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Stroke
Keywords: Stroke; Early Ambulation; Rehabilitation; Physical Therapy; Randomized controlled trial
MeSH Terms: conditions — Stroke | interventions — Early Ambulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early mobilization (Experimental): The Intervention Group - Early Mobilization - will follow the early physiotherapy program within the first 24 - 48 hours after stroke, five times per week for 30 plus a time spent out of bed (sitting).
  Interventions: Other: Early mobilization
- Control (No Intervention): The Control Group will follow within the routines of the hospital as is usually done.

INTERVENTIONS:
Other: Early mobilization — The Intervention Group - Early Mobilization - will follow the early physiotherapy program within the first 24 - 48 hours after acute ischemic stroke, five times per week for 30 minutes plus time to spent out of bed (sitting).
  Other Names: Early Physiotherapy Program
  Arms: Early mobilization

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a rehabilitation (physiotherapy) program in patients with acute ischemic stroke in Acute Vascular Unit and in general ward of Hospital de Clínicas de Porto Alegre, and to verify the degree of disability at fourteenth and third month, functional improvement at third month, the frequency of deaths and incidence of complications due to immobility and quantify the time spent in hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of acute ischemic stroke (first or recurrent) confirmed by CCT or MRI admitted to the Acute Vascular Unit of HCPA between the first 48 hours of onset of symptoms.
* Patients older than 18 years.
* Patients clinically and hemodynamically stable (SBP 120-220 mmHg, SatO2 up to 92% with or without supplementation, HR between 60 and 100 bmp, body temperature below 38 and RR below 25 bpm).
* Patients are able to react to verbal commands even without being fully alert (Glasgow Scale above 8).
* Prior Rankin until 3
* Motor deficit and / or coordination measured by the NIHSS

Exclusion Criteria:

* Patients with clinical and / or hemodynamic instability
* Patients with hemorrhagic stroke or TIA (transient ischemic attack).
* Patients with progressive neurological disease and acute coronary disease and / or unstable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-12 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Disability | three months
  Outcome measure are assessed by Modified Rankin Scale. Good outcome was predefined as an mRS score of 0 to 2 and poor outcome of 3 to 6.

SECONDARY OUTCOMES:
Minimum or no Disability | three months
  Measured by the modified Ranking Scale with score of 0 to 1.
Independence in activities of daily living | three months
  Measured by the modified Barthel Index, where score < 75 indicate dependence and score > 75 is independence.
Long of stay at hospital | three month
  Number of days in hospital
Death | three month
  Determined by a blinded review of the clinical details by the investigators.
Incidence of complications | three month
  Number of complications (pneumonia and deep vein thrombosis) at three month

CONTACTS AND LOCATIONS:
Overall Officials: Sheila CO Martins, Physician, Principal Investigator — Hospital de Clínicas de Porto Alegre (Hospital)
Locations (1):
- Hospital de Clínicas de Porto Alegre (Hospital), Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Clark B, Whitall J, Kwakkel G, Mehrholz J, Ewings S, Burridge J. The effect of time spent in rehabilitation on activity limitation and impairment after stroke. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD012612. doi: 10.1002/14651858.CD012612.pub2. PMID 34695300